CLINICAL TRIAL: NCT06238752
Title: First-line Apatinib Combined With Tislelizumab and Chemotherapy for Advanced Gastric and Gastroesophageal Junction(G/GEJ) Adenocarcinoma Patients With Poor Prognosis: A Prospective Exploratory Study
Brief Title: First-line Apatinib Combined With Tislelizumab and Chemotherapy for Advanced GC
Acronym: RENMIN-213
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Yongshun Chen, prof, Renmin Hospital of Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WDRY2022-K097
Record Dates: First submitted 2024-01-24; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Advanced Gastric Adenocarcinoma
Keywords: Apatinib; Tislelizumab; Chemotherapy; Advanced; Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — tislelizumab; Drug Therapy; Psychotherapy, Multiple

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- first-line treatment with the combination of apatinib, immune checkpoint inhibitor and chemotherapy (Experimental): Patients received 8 cycles of apatinib (250 mg, qd, d1-14), tislelizumab(200 mg d1), and oxaliplatin (130 mg/m2, d1) plus oral capecitabine (1000 mg/m2, bid, d1-14) every 3 weeks, with a maintenance therapy with apatinib plus tislelizumab for a maximum of 1 year. Homogeneous patients receiving ICIs combined with chemotherapy at the same time were deemed as the control group for efficacy.
  Interventions: Drug: Apatinib Combined With Tislelizumab and Chemotherapy

INTERVENTIONS:
Drug: Apatinib Combined With Tislelizumab and Chemotherapy — apatinib (250 mg, qd, d1-14), tislelizumab(200 mg d1), and oxaliplatin (130 mg/m2, d1) plus oral capecitabine (1000 mg/m2, bid, d1-14) every 3 weeks
  Other Names: Combined therapy

SUMMARY:
In this clinical study, investigators explore the efficacy and safety of a combination therapy regimen with antiangiogenic agent (apatinib), ICI (tislelizumab), and chemotherapy (capecitabine+ Oxaliplatin, XELOX) as first-line treatment for HER2-negative, advanced G/GEJ cancer patients with signet ring cell carcinoma or peritoneal metastasis.

DETAILED DESCRIPTION:
Patients received 8 cycles of apatinib (250 mg, qd, d1-14), tislelizumab (200 mg d1), and oxaliplatin (130 mg/m2, d1) plus oral capecitabine (1000 mg/m2, bid, d1-14) every 3 weeks, with a maintenance therapy with apatinib plus tislelizumab for a maximum of 1 year. Homogeneous patients receiving ICIs combined with chemotherapy at the same time were deemed as the control group for efficacy.

ELIGIBILITY:
Inclusion Criteria:After providing written consent before participation in the study, patients must fulfill all of the following criteria. If a subject is found not to meet any of the following criteria before the first dose of the therapy regimen, the subject will not be started on the study treatment but will be withdrawn from the study.

1. Sex: Men and women
2. Age (at the time of informed consent): 18 years and older
3. Patients with unresectable advanced or recurrent gastric cancer (including esophagogastric junction cancer) that has been istologically confirmed to be adenocarcinoma and has not been treated with the first-line therapy with systemic antitumor agents for advanced or recurrent gastric cancer (including esophagogastric junction cancer).For patients who have received neoadjuvant or adjuvant chemotherapy (including chemoradiotherapy) in combination with curative or endoscopic surgery (R0 resection confirmed), the chemotherapy in the last regimen must be completed by at least 180 days before the date of recurrence.
4. Have at least one measurable lesion, as defined in the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1), on computed tomography (CT) or magnetic resonance imaging (MRI) within 28 days before enrolled in the study
5. Able to provide tumor tissue specimens (archival or fresh biopsy specimens) for PD-L1 expression analysis. For patients who are unable to undergo another biopsy, archival specimens may be used as an alternative.
6. ECOG PS score 0 or 1
7. Have a life expectancy of at least 3 months
8. Have latest laboratory data meeting the criteria below within 7 days before enrolled. If the date of the laboratory tests at enrolled is not within 7 days before the first dose of the therapy regimen, testing should be repeated within 7 days before the first dose of the therapy regimen, and the latest laboratory data before the first dose of the therapy regimen must be confirmed to meet the following criteria. Moreover, laboratory data will not be valid if the patient has received a granulocyte colony stimulating factor (G-CSF) or blood transfusion within 14 days before testing.

   * White blood cells ≥3000 cells per μL, and neutrophil count ≥1000 cells per μL
   * Platelets ≥70 000 per μL
   * haemoglobin ≥80 g/L
   * Aspartate aminotransferase (AST) and alanine aminotransferase ≤3 times the limit of normal (ULN) or ≤5 times the ULN in patients with liver metastases
   * Total bilirubin ≤1.5 times the ULN
   * International Normalized Ratio (INR) ≤1.5
   * Creatinine ≤1.5 times the ULN or creatinine clearance >30 mL/min
   * albumin ≥3g/L
9. Women of childbearing potential (including women with chemical menopause or no menstruation for other medical reasons) must agree to use contraception from the time of informed consent until at least 5 months after the last dose of the therapy regimen, whichever comes later. Also, women must agree not to breastfeed from the time of informed consent until at least 5 months after the last dose of the therapy regimen, whichever comes later.
10. Men must agree to use contraception from the start of the study treatment until at least 7 months after the last dose of the therapy regimen.

Exclusion Criteria:Patients meeting any of the following criteria at assessment for participation will be excluded from the study. If a randomized subject is found to meet any of the following criteria before the first dose of the therapy regimen, the subject will not be started on the study treatment but will be withdrawn from the study.

1. Patients with HER2-positive or indeterminate gastric cancer (Determination for positive is made on the basis of the reference in each site. If there is no reference, rough indication for positive is 3+ by immunohistochemistry [IHC], or 2+ by IHC and positive by in situ hybridization [ISH]).
2. multiple cancers (with the exception of completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, and superficial bladder cancer, and any other cancers that have not recurred for at least 5 years)
3. previous treatment with ICIs, chemotherapy or anti-angiogenic drug
4. interstitial lung disease or pulmonary fibrosis
5. Have concurrent autoimmune disease or a history of chronic or recurrent autoimmune disease. Patients with Type 1 diabetes mellitus, hypothyroidism which is manageable by hormone replacement or skin disorders not requiring systemic treatment (such as vitiligo, psoriasis, or alopecia) are permitted to be enrolled.
6. Unable to take oral medicines
7. Have a current or past history of severe hypersensitivity to any other antibody products
8. Have concurrent diverticulitis or symptomatic gastrointestinal ulcerative disease
9. Have experienced a transient ischemic attack, cerebrovascular accident, thrombosis or thromboembolism (pulmonary arterial embolism or deep vein thrombosis) within 180 days before enrolled
10. Have a history of uncontrollable or significant cardiovascular disease meeting any of the following;

    * myocardial infarction within 180 days before randomization
    * uncontrollable angina pectoris within 180 days before randomization
    * arrhythmia requiring treatment
11. Are receiving or require anticoagulant therapy (other than antiplatelet therapy including low dose aspirin) for a disease
12. Have uncontrollable diabetes mellitus
13. Have systemic infection requiring treatment
14. Are contraindicated for oxaliplatin, capecitabine, tislelizumab, apatinib
15. Have received radiotherapy for gastric cancer within 28 days before randomization or radiotherapy for bone metastases within 14 days before randomization
16. Have received any radiopharmaceuticals (except for examination or diagnostic use of radiopharmaceuticals) within 56 days before randomization
17. Have a positive test result for human immunodeficiency virus-1 (HIV-1) antibody, human immunodeficiency virus-2 (HIV-2) antibody, human T-lymphotropic virus-1 (HTLV-1) antibody, hepatitis B surface protein (HBs) antigen, or hepatitis C virus (HCV) antibody
18. Are pregnant or breastfeeding, or possibly pregnant
19. Have received any other unapproved drug (e.g., marketed drugs unapproved for gastric cancer, investigational use of drugs, unapproved combined formulations, unapproved dosage forms) within 28 days (or within 90 days for antibody products) before enrolled
20. With peripheral neuropathy of Grade ≥2
21. severe symptoms (including a rapid decline in ECOG performance; rapidly worsening symptoms; requiring urgent medical intervention), or active systemic infection, blood clotting disorder or other active major disease
22. Are incapable of providing consent for specific reasons, such as concurrent dementia
23. Are otherwise inappropriate for this study in the investigator's opinion.
24. Have received a live/attenuated vaccine within 28 days before randomization untreated central nervous system metastases peripheral neuropathy (> grade 1), known history of positive test for human immunodeficiency virus or known acquired immunodeficiency syndrome, concurrent diverticulitis or symptomatic gastrointestinal ulcerative disease, severe symptoms (including a rapid decline in ECOG performance; rapidly worsening symptoms; requiring urgent medical intervention), or active systemic infection, blood clotting disorder or other active major disease were excluded from the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
PFS | through study completion, an average of 1 year
  progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Chen, Study Chair — Renmin Hospital of Wuhan University
Locations (1):
- Renmin hosptial of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Open to researchers who need it
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication
Access Criteria: yongshun2007@163.com